CLINICAL TRIAL: NCT00685698
Title: An Open-Label, Single-Arm, Multi-Center Study of TG-873870 for Treating Patients With Diabetic Foot Infections of Mild to Moderate Severity Associated With Gram-Positive Pathogens
Brief Title: Safety and Efficacy Study of TG-873870 (Nemonoxacin) in Diabetic Foot Infections
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: TaiGen Biotechnology Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: TG-873870-04
Record Dates: First submitted 2008-05-22; First posted 2008-05-28 (Estimated); Results first posted 2015-01-09 (Estimated); Last update posted 2025-07-01 (Actual); Status verified 2014-12

CONDITIONS: Diabetic Foot Infections
Keywords: Diabetic Foot Infections, DFI, Nemonoxacin
MeSH Terms: interventions — nemonoxacin

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Nemonoxacin (Other): Nemonoxacin 750 mg,oral administration, single-arm, once daily 7±1 and 14±1 days.
  Interventions: Drug: TG-873870 (Nemonoxacin)

INTERVENTIONS:
Drug: TG-873870 (Nemonoxacin) — 750 mg
  Other Names: Taigexyn

SUMMARY:
Safety and Efficacy Study of TG-873870 (Nemonoxacin) in Diabetic Foot Infections

DETAILED DESCRIPTION:
This study will assess the safety and efficacy of TG-873870 (Nemonoxacin) in patients with Diabetic Foot Infections. Pharmacokinetic (PK) and pharmacodynamic (PD) assessment will be conducted in a subgroup of eight consenting patients.

ELIGIBILITY:
Inclusion Criteria:

* Body weight ≥ 40 kg
* Previously known or newly diagnosed diabetes mellitus, including type 1 and type 2 (per the American Diabetes Association guidelines), which is controlled by proper lifestyle (diet, exercise) or treatment with either oral medications or insulin
* Patients' HbA1c ≦ 12% at screening
* Clinically defined diabetic foot infection of mild or moderate severity (PEDIS grade 2-3) as based on the guideline of the Infectious Diseases Society of America. It includes any inframalleolar infection of the soft-tissue, such as paronychia, cellulitis, myositis, abscesses, and tendonitis
* Evidence of necrotic tissue, purulent collections or abscess that may require excision, incision or drainage (based on investigator's judgment, and a surgeon if needed)
* Must be able to provide suitable tissue specimens (preferably obtained by biopsy or tissue curettage, or purulent fluid aspiration, rather than by swabbing) from the infected wound (after appropriate cleansing and debridement) for Gram-staining and bacterial cultures (aerobes and anaerobes)
* A confirmed Gram-positive pathogen infection by Gram-stain. The criterion to determine patient's eligibility for study recruitment is a Gram-stained smear with at least 1 Gram-positive organism seen in at least two high power fields. A solely Gram-positive pathogen infection or a polymicrobial infection including Gram-positive and Gram-negative pathogens are acceptable within the framework of the study

Exclusion Criteria:

* A co-morbid disease condition that could compromise evaluation or participation in this study, such as severe hepatic disease (e.g., active hepatitis, decompensated liver cirrhosis), renal failure (estimated creatinine clearance [CrCl] <30 ml/minute or need for hemodialysis or peritoneal dialysis), or active systemic malignancy (advanced or metastatic), unless enrollment is deemed appropriate at the discretion of the Investigator with prior consultation with the study Medical Monitor
* History of prolonged QTc interval or a medical condition requiring the use of a concomitant medication that is associated with an increased QTc interval (e.g., class I or class III anti-arrhythmic agents)
* Contact dermatitis over the infected skin area, infected third-degree burn wounds, necrotizing fascitis, extensive gangrene, pyoderma gangrenosum, deep vein thrombosis, shock, or any medical disorder that could either interfere with the evaluation of treatment or the response of the patient to therapy
* Radiological evidence of bone or joints infection within 7 days prior to or at screening, i.e. potential osteomyelitis or septic arthritis
* Clinically defined uninfected or severe infection (PEDIS grade 1 or 4) as based on the Infectious Diseases Society of America classification system
* Any known severe immunosuppressive condition, such as an active hematological malignancy, HIV infection or active treatment with any immunosuppressive drug (including corticosteroids at a dose of >20 mg/day of prednisone, or its equivalent)
* Has received or will be receiving chemotherapy or oncolytics within six months prior to entering or during the study
* History of current or active alcohol abuse (>3 drinks daily or binge drinking) or any illicit drug use
* Known or suspected critical ischemia of the affected limb (based on investigators' clinical judgments and vascular assessment)
* Wound that contains or is proximate to any prosthetic materials or devices that is/are not scheduled for removal
* Patient with a foot infection that, in the investigator's judgment, is severe enough to require hospitalization or intravenous antibiotic therapy
* Neutrophil count <1000 cells/mm3

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Actual)
Dates: Start 2008-06; Primary Completion 2009-04 (Actual); Study Completion 2009-06 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Kuang-Chung Shih, M.D., Study Chair — Tri-Service General Hospital, Taipei, Taiwan; Jawl-Shan Hwang, M.D., Principal Investigator — Cheng-Gung Memorial Hospital - LinKou, Taiwan; Te-Lin Hsia, M.D., Principal Investigator — Cardinal Tien Hospital (CTH), Taiwan; Jung-Fu Chen, M.D., Principal Investigator — Chang Gung Memorial Hospital- Kaoshiung, Taiwan; Chien-Wen Chou, M.D., Principal Investigator — Chi-Mei Medical Center, Tainan, Taiwan; Che-Han Hsu, M.D., Principal Investigator — Cheng Ching Hospital, Taichung, Taiwan; Joseph De Santo, M.D., Principal Investigator — HealthCare Partners, Pasadena, USA; Lee Rogers, M.D., Principal Investigator — The Amputation Prevention Center at Broadlawns Medical Center, Des Moines, USA; Kwei Quartey, M.D., Principal Investigator — HealthCare Partners, Montebello, USA; Lynn Tudhope, M.D., Principal Investigator — Montana Hospital, Pretoria, South Africa; Andre Tudhope, M.D., Principal Investigator — Jubilee Clinical Trial Center, Hammanskraal, South Africa; Mohammed Fulat, M.D., Principal Investigator — Eastmed Academic Clinical Trial Center, East Lynne, South Africa; Dirkie van Rensburg, M.D., Principal Investigator — Park Medical Center, Witbank, South Africa; Mashra Gani, M.D., Principal Investigator — Mercantile Clinical Trial Center, Korsten, South Africa; Piroon Mootsitkapun, M.D., Principal Investigator — Faculty of Medicine, Khon Kaen University, Thailand; Chieh-Feng Chen, M.D., Principal Investigator — Wan Fang Hospital, Taipei, Taiwan
Locations (16):
- United States (3):
  - HealthCare Partners, Montebello, California
  - HealthCare Partners, Pasadena, California
  - The Amputation Prevention Center at Broadlawns Medical Center, Des Moines, Iowa
- South Africa (5):
  - Eastmed Academic Clinical Trial Center, East Lynne, Gauteng
  - Jubilee Clinical Trial Center, Hammanskraal, Gauteng
  - Montana Hospital, Pretoria, Gauteng
  - Park Medical Center, Witbank, Gauteng
  - Mercantile Clinical Trial Center, Korsten, Port Elizabeth
- Taiwan (7):
  - Chang Gung Memorial Hospital- Kaoshiung, Taiwan, Kaohsiung City
  - Cheng Ching Hospital, Taichung, Taiwan, Taichung
  - Chi-Mei Medical Center, Tainan, Taiwan, Tainan
  - Cardinal Tien Hospital (CTH), Taiwan, Taipei
  - Tri-Service General Hospital, Taipei, Taiwan, Taipei
  - Wan Fang Hospital, Taipei
  - Cheng-Gung Memorial Hospital - LinKou, Taiwan, Taoyuan District
- Faculty of Medicine, Khon Kaen University, Khon Kaen, Thailand

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Patients were assessed during the 1- to 2-day screening phase (Visit 1) to determine their eligibility. Eligible patients demonstrating the presence of at least one Gram-positive organism on the basis of Gram-stain could begin treatment with study medication the same day (Day 1, Visit 1).
Period: Overall Study
Arm/Group | Nemonoxacin
Started | 38
Completed | 25
Not Completed | 13
Not completed — Withdrawal by Subject | 1
Not completed — Protocol Violation | 6
Not completed — Adverse Event | 3
Not completed — CULTURE GRAM NEG SPECIES | 1
Not completed — CULTURE RESULTS: GRAM-VE | 1
Not completed — NO GRAM POSITIVE CULTURE GROWN | 1

BASELINE CHARACTERISTICS:
Population: The ITT population consists of all patients from the Enrolled population who took at least one whole dose of study medication (three capsules) and who exhibited at least one Gram-positive pathogen at Baseline (Visit 1) as confirmed by culture of wound tissue by the central (or local) laboratory.
Arm/Group | Nemonoxacin
Number analyzed (Participants) | 33
Age, Continuous [Mean (Standard Deviation); unit: years] | 59.2 (11.87)
Age, Continuous [Median (Full Range); unit: years] | 57.0 [39 to 87]
Age, Customized [Number; unit: participants]
  < 20 years | 0
  >= 20 and < 30 years | 0
  >= 30 and < 40 years | 1
  >= 40 and < 50 years | 8
  >= 50 and < 60 years | 11
  >= 60 and < 70 years | 3
  >= 70 and < 80 years | 9
  >= 80 years | 1
Sex: Female, Male [Count of Participants; unit: Participants] — Most patients (66.7%) were male.
  Participants
    Female | 11
    Male | 22
Race/Ethnicity, Customized [Number; unit: participants] — Most patients (45.5%) were white.
  participants
    White | 15
    Black | 7
    Asian | 5
    Native Hawaiian or Other Pacific Islander | 0
    American Indian or Alaska Native | 0
    Other | 6
Type of Diabetes [Number; unit: participants] — Most patients (90.9%) were type 2 diabetes.
  participants
    Type 1 (Juvenile Onset) | 3
    Type 2 (Adult Onset) | 30
Time Since Diabetes Diagnosis [Mean (Standard Deviation); unit: years] | 8.0 (6.49)
Distribution of Time Since Diabetes Diagnosis [Number; unit: participants]
  < 5 years | 12
  >= 5 and < 10 years | 8
  >= 10 and < 20 years | 9
  >= 20 and < 30 years | 2
  >= 30 and < 40 years | 0
  >= 40 years | 0
  Missing | 2
Most Recent HbA1c % Result [Number; unit: participants] — Performed within 6 Months prior to Visit 1.
  participants
    < 6.5% | 2
    >= 6.5% and < 7.0% | 3
    >= 7.0% and < 9.0% | 10
    >= 9.0% and < 10.0% | 3
    >= 10.0% and < 11.0% | 2
    >= 11.0% and < 12.0% | 1
    >= 12.0% | 0
    Missing | 12
HbA1c % Result at Visit 1 [Number; unit: participants] — Central Laboratory Data if available. Local Laboratory Data if not available. Most patients (54.5%) had a baseline HbA1c value between 7.0 and 9.0%, and 24.2% (8/33) appeared to be well controlled with values below 7.0%.
  participants
    < 6.5% | 6
    >= 6.5% and < 7.0% | 2
    >= 7.0% and < 9.0% | 18
    >= 9.0% and < 10.0% | 3
    >= 10.0% and < 11.0% | 1
    >= 11.0% and < 12.0% | 2
    >= 12.0% | 1
Current treatment for Diabetes [Number; unit: participants] — Most patients (75.8%) received oral agent(s) for their treatment of diabetes, and nearly half the patients were on insulin.
  participants
    Diet and Exercise | 20
    Oral Agent | 25
    Insulin | 16
Time Since Diabetes Diagnosis [Median (Full Range); unit: years] — The patient population included some newly diagnosed individuals.
  years | 6.0 [0 to 23]

OUTCOME MEASURES:

1. Primary Outcome: Clinical Success (in ITT Population)
Description: Clinical Success
  * Resolution is defined as total resolution of all pretreatment clinically significant signs and symptoms of infection and no development of any systemic evidence of infection.
  * Improvement is defined as resolution of more than two, but not all, pretreatment clinical signs and symptoms, or partial resolution of all clinical signs and symptoms relative to the baseline assessment, with no further need for antibiotic therapy, and no need for infection-related surgical interventions.
Time Frame: Test of Cure Visit, 12±2 days after End of Treatment Visit/Early Termination
Population: All eligible patients who took at least one whole dose of study drug and had at least 1 gram-positive pathogen identified at the Baseline Visit (Visit 1).
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Nemonoxacin
Number analyzed (Participants) | 33
percentage of participants | 95.7 [78.1 to 99.9]

2. Secondary Outcome: Microbiological Success Rate
Description: Microbiological Success
  * Eradicated, defined as absence of the original pathogen(s) from a repeat culture of the original infection site performed at the TOC visit.
  * Presumed Eradicated, defined as meeting the definition for Clinical Success at the TOC visit, but tissue sample could be obtained for culture from the original infection site.
    * TOC=Test of Cure
Time Frame: Test of Cure Visit, 12±2 days after End of Treatment Visit/Early Termination
Measure: Number (95% Confidence Interval); unit: percentage of participants
Groups:
- Nemonoxacin (ITT Population at Test of Cure Visit); Nemonoxacin (PP Population at Test of Cure Visit): Nemonoxacin 750 mg,oral administration, single-arm, once daily 7±1 and 14±1 days.
  TG-873870 (Nemonoxacin): 750 mg
Arm/Group | Nemonoxacin (ITT Population at Test of Cure Visit) | Nemonoxacin (PP Population at Test of Cure Visit)
Number analyzed (Participants) | 33 | 20
percentage of participants | 82.6 [61.2 to 95.0] | 89.5 [66.9 to 98.7]

3. Secondary Outcome: Clinical Success (in PP Population)
Description: as for outcome 1
Time Frame: Test of Cure Visit, 12±2 days after End of Treatment Visit/Early Termination
Population: All eligible patients who took at least one whole dose of study drug and had at least 1 gram-positive pathogen identified at the Baseline Visit (Visit 1), and adhered to the protocol without major protocol violations.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Nemonoxacin
Number analyzed (Participants) | 20
percentage of participants | 94.7 [74.0 to 99.9]

4. Secondary Outcome: Clinical Success (at End of Treatment/Early Termination)
Description: as for outcome 1
Time Frame: End of Treatment/Early Termination Visit; 7±1, 14±1, 21±1 or 28±1 days after Baseline (Day 1)
Measure: Number (95% Confidence Interval); unit: percentage of participants
Groups:
- Nemonoxacin (ITT Population at EOT/ET); Nemonoxacin (PP Population at EOT/ET): Nemonoxacin 750 mg,oral administration, single-arm, once daily 7±1 and 14±1 days.
  TG-873870 (Nemonoxacin): 750 mg
Arm/Group | Nemonoxacin (ITT Population at EOT/ET) | Nemonoxacin (PP Population at EOT/ET)
Number analyzed (Participants) | 33 | 24
percentage of participants | 100.0 [87.7 to 100.0] | 100.0 [85.2 to 100.0]

5. Secondary Outcome: Per-Pathogen Clinical Responses (at Test of Cure)
Description: Clinical responses were assessed on a per-pathogen basis for the most frequently isolated pathogens at baseline (i.e., present in four or more patients), including MRSA. Clinical Responses were assessed at Test of Cure visit within each of the ITT and PP populations. Insufficient numbers prevented reporting Clinical Success rates for Streptococcus pyogenes in the PP population.
Time Frame: Test of Cure Visit, 12±2 days after End of Treatment Visit/Early Termination
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Nemonoxacin (ITT Population at Test of Cure Visit) | Nemonoxacin (PP Population at Test of Cure Visit)
Number analyzed (Participants) | 33 | 20
percentage of participants
  Staphylococcus aureus | 100.0 [78.2 to 100.0] | 100.0 [73.5 to 100.0]
  Escherichia coli (in ITT population) | 100.0 [54.1 to 100.0] | 100.0 [39.8 to 100.0]
  Enterococcus faecalis (in ITT population) | 100.0 [39.8 to 100.0] | 100.0 [39.8 to 100.0]
  Streptococcus agalactiae (in ITT population) | 100.0 [29.2 to 100.0] | 100.0 [29.2 to 100.0]
  Streptococcus pyogenes (in ITT population) | 100.0 [39.8 to 100.0] | NA [NA to NA] — Insufficient numbers prevented reporting Clinical Success rate for Streptococcus pyogenes in the PP population.

6. Secondary Outcome: Per-Pathogen Clinical Response (at End of Treatment/Early Termination)
Description: Clinical responses were assessed on a per-pathogen basis for the most frequently isolated pathogens at baseline (i.e., present in four or more patients), including MRSA. Clinical Responses were assessed at at End of Treatment/Early Termination within each of the ITT and PP populations. Insufficient numbers prevented reporting Clinical Success rates for Streptococcus pyogenes in the PP population.
Time Frame: End of Treatment/Early Termination Visit; 7±1, 14±1, 21±1 or 28±1 days after Baseline (Day 1)
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Nemonoxacin (ITT Population at EOT/ET) | Nemonoxacin (PP Population at EOT/ET)
Number analyzed (Participants) | 33 | 24
percentage of participants
  Staphylococcus aureus (in ITT population) | 100.0 [81.5 to 100.0] | 100.0 [78.2 to 100.0]
  Escherichia coli (in ITT population) | 100.0 [54.1 to 100.0] | 100.0 [39.8 to 100.0]
  Enterococcus faecalis (in ITT population) | 100.0 [47.8 to 100.0] | 100.0 [47.8 to 100.0]
  Streptococcus agalactiae (in ITT population) | 100.0 [39.8 to 100.0] | 100.0 [29.2 to 100.0]
  Streptococcus pyogenes (in ITT population) | 100.0 [39.8 to 100.0] | NA [NA to NA] — Insufficient numbers prevented reporting Clinical Success rate for Streptococcus pyogenes in the PP population.

7. Secondary Outcome: Per-Pathogen Microbiological Responses
Description: Microbiological responses were assessed on a per-pathogen basis for the most frequently isolated pathogens at baseline (i.e., present in four or more patients), including MRSA. Microbiological Responses were assessed at Test of Cure visit within each of the ITT and PP populations. Insufficient numbers prevented reporting Microbiological Success rates for Streptococcus pyogenes in the PP population.
Time Frame: Test of Cure Visit, 12±2 days after End of Treatment Visit/Early Termination
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Nemonoxacin (ITT Population at Test of Cure Visit) | Nemonoxacin (PP Population at Test of Cure Visit)
Number analyzed (Participants) | 33 | 20
percentage of participants
  Staphylococcus aureus (in ITT population) | 93.3 [68.1 to 99.8] | 100.0 [73.5 to 100.0]
  Escherichia coli (in ITT population) | 66.7 [22.3 to 95.7] | 75.0 [19.4 to 99.4]
  Enterococcus faecalis (in ITT population) | 75.0 [19.4 to 99.4] | 75.0 [19.4 to 99.4]
  Streptococcus agalactiae (in ITT population) | 100.0 [29.2 to 100.0] | 100.0 [29.2 to 100.0]
  Streptococcus pyogenes (in ITT population) | 100.0 [39.8 to 100.0] | NA [NA to NA] — Insufficient numbers prevented reporting Microbiological Success rate for Streptococcus pyogenes in the PP population.

8. Secondary Outcome: Total Wound Score (at Test of Cure in ITT Population)
Description: The Diabetic Foot Infection (DFI) Wound Scores will be used to evaluate the wound assessment at baseline and Test of Cure visits. The wound composite score was based on combining the general wound parameters (signs and symptoms of infection), and wound measurements (length, width, depth). Each wound parameter was assigned a score based on severity, with higher scores defining greater severity. For wound measurements and undermining, larger measurements received higher scores. The minimum and maximum score are 3 and 49, respectively.
Time Frame: Visit 1 (Baseline); Test of Cure Visit, 12±2 days after End of Treatment Visit/Early Termination
Measure: Mean (Standard Deviation); unit: scores on a scale
Groups:
- Nemonoxacin (at Baseline, ITT Population); Nemonoxacin (at Test of Cure Visit, ITT Population); Nemonoxacin (Change From Baseline to Test of Cure Visit): Nemonoxacin 750 mg,oral administration, single-arm, once daily 7±1 and 14±1 days.
  TG-873870 (Nemonoxacin): 750 mg
Arm/Group | Nemonoxacin (at Baseline, ITT Population) | Nemonoxacin (at Test of Cure Visit, ITT Population) | Nemonoxacin (Change From Baseline to Test of Cure Visit)
Number analyzed (Participants) | 33 | 28 | 28
scores on a scale | 16.9 (6.30) | 6.0 (3.67) | -11.2 (6.91)

9. Secondary Outcome: Total Wound Score (at Test of Cure in PP Population)
Description: as for outcome 8
Time Frame: Visit 1 (Baseline); Test of Cure Visit, 12±2 days after End of Treatment Visit/Early Termination
Measure: Mean (Standard Deviation); unit: scores on a scale
Groups:
- Nemonoxacin (at Baseline, PP Population); Nemonoxacin (at Test of Cure Visit, PP Population); Nemonoxacin (Change From Baseline to Test of Cure Visit): Nemonoxacin 750 mg,oral administration, single-arm, once daily 7±1 and 14±1 days.
  TG-873870 (Nemonoxacin): 750 mg
Arm/Group | Nemonoxacin (at Baseline, PP Population) | Nemonoxacin (at Test of Cure Visit, PP Population) | Nemonoxacin (Change From Baseline to Test of Cure Visit)
Number analyzed (Participants) | 20 | 19 | 19
scores on a scale | 18.2 (6.54) | 5.0 (2.79) | -12.9 (7.10)

10. Secondary Outcome: Total Wound Score (at End of Treatment/ Early Termination in ITT Population)
Description: The Diabetic Foot Infection (DFI) Wound Scores will be used to evaluate the wound assessment at baseline and End of Treatment/ Early Termination visits. The wound composite score was based on combining the general wound parameters (signs and symptoms of infection), and wound measurements (length, width, depth). Each wound parameter was assigned a score based on severity, with higher scores defining greater severity. For wound measurements and undermining, larger measurements received higher scores. The minimum and maximum score are 3 and 49, respectively.
Time Frame: Visit 1 (Baseline); End of Treatment/Early Termination Visit; 7±1, 14±1, 21±1 or 28±1 days after Baseline (Day 1)
Measure: Mean (Standard Deviation); unit: scores on a scale
Groups:
- Nemonoxacin (at EOT/ET Visit, ITT Population); Nemonoxacin (Change From Baseline to EOT/ET Visit): Nemonoxacin 750 mg,oral administration, single-arm, once daily 7±1 and 14±1 days.
  TG-873870 (Nemonoxacin): 750 mg
Arm/Group | Nemonoxacin (at Baseline, ITT Population) | Nemonoxacin (at EOT/ET Visit, ITT Population) | Nemonoxacin (Change From Baseline to EOT/ET Visit)
Number analyzed (Participants) | 33 | 32 | 32
scores on a scale | 16.9 (6.30) | 7.2 (4.65) | -9.6 (6.35)

11. Secondary Outcome: Total Wound Score (at End of Treatment/ Early Termination in PP Population)
Description: as for outcome 8
Time Frame: Visit 1 (Baseline); End of Treatment/Early Termination Visit; 7±1, 14±1, 21±1 or 28±1 days after Baseline (Day 1)
Measure: Mean (Standard Deviation); unit: scores on a scale
Groups:
- Nemonoxacin (at EOT/ET Visit, PP Population); Nemonoxacin (Change From Baseline to EOT/ET Visit): Nemonoxacin 750 mg,oral administration, single-arm, once daily 7±1 and 14±1 days.
  TG-873870 (Nemonoxacin): 750 mg
Arm/Group | Nemonoxacin (at Baseline, PP Population) | Nemonoxacin (at EOT/ET Visit, PP Population) | Nemonoxacin (Change From Baseline to EOT/ET Visit)
Number analyzed (Participants) | 20 | 20 | 20
scores on a scale | 18.2 (6.54) | 6.2 (4.31) | -12.1 (6.44)

12. Secondary Outcome: Diabetic Foot Assessment (PEDIS) Shifts From Baseline at End of Treatment/Early Termination in ITT Population
Description: The number of patients within each of the PEDIS grading categories (uninfected, mild, moderate and severe) at baseline and End of Treatment/Early Termination.
Time Frame: End of Treatment/Early Termination Visit; 7±1, 14±1, 21±1 or 28±1 days after Baseline (Day 1)
Measure: Number; unit: participants
Arm/Group | Nemonoxacin
Number analyzed (Participants) | 33
participants
  Uninfected to Uninfected | 0
  Uninfected to Mild | 0
  Uninfected to Moderate | 0
  Uninfected to Severe | 0
  Mild to Uninfected | 8
  Mild to Mild | 4
  Mild to Moderate | 0
  Mild to Severe | 0
  Moderate to Uninfected | 12
  Moderate to Mild | 5
  Moderate to Moderate | 3
  Moderate to Severe | 0
  Severe to Uninfected | 0
  Severe to Mild | 0
  Severe to Moderate | 0
  Severe to Severe | 0

13. Secondary Outcome: Diabetic Foot Assessment (PEDIS) Shifts From Baseline at Test of Cure in ITT Population
Description: The number of patients within each of the PEDIS grading categories (uninfected, mild, moderate and severe) at baseline and Test of Cure.
Time Frame: Test of Cure Visit, 12±2 days after End of Treatment Visit/Early Termination
Measure: Number; unit: participants
Arm/Group | Nemonoxacin
Number analyzed (Participants) | 33
participants
  Uninfected to Uninfected | 0
  Uninfected to Mild | 0
  Uninfected to Moderate | 0
  Uninfected to Severe | 0
  Mild to Uninfected | 8
  Mild to Mild | 2
  Mild to Moderate | 0
  Mild to Severe | 0
  Moderate to Uninfected | 15
  Moderate to Mild | 3
  Moderate to Moderate | 0
  Moderate to Severe | 0
  Severe to Uninfected | 0
  Severe to Mild | 0
  Severe to Moderate | 0
  Severe to Severe | 0

14. Secondary Outcome: Diabetic Foot Assessment (PEDIS) Shifts From Baseline at End of Treatment/Early Termination in PP Population
Description: as for outcome 12
Time Frame: End of Treatment/Early Termination Visit; 7±1, 14±1, 21±1 or 28±1 days after Baseline (Day 1)
Measure: Number; unit: participants
Arm/Group | Nemonoxacin
Number analyzed (Participants) | 20
participants
  Uninfected to Uninfected | 0
  Uninfected to Mild | 0
  Uninfected to Moderate | 0
  Uninfected to Severe | 0
  Mild to Uninfected | 6
  Mild to Mild | 1
  Mild to Moderate | 0
  Mild to Severe | 0
  Moderate to Uninfected | 9
  Moderate to Mild | 2
  Moderate to Moderate | 2
  Moderate to Severe | 0
  Severe to Uninfected | 0
  Severe to Mild | 0
  Severe to Moderate | 0
  Severe to Severe | 0

15. Secondary Outcome: Diabetic Foot Assessment (PEDIS) Shifts From Baseline at Test of Cure in PP Population
Description: as for outcome 13
Time Frame: Test of Cure Visit, 12±2 days after End of Treatment Visit/Early Termination
Measure: Number; unit: participants
Arm/Group | Nemonoxacin
Number analyzed (Participants) | 20
participants
  Uninfected to Uninfected | 0
  Uninfected to Mild | 0
  Uninfected to Moderate | 0
  Uninfected to Severe | 0
  Mild to Uninfected | 6
  Mild to Mild | 1
  Mild to Moderate | 0
  Mild to Severe | 0
  Moderate to Uninfected | 11
  Moderate to Mild | 1
  Moderate to Moderate | 0
  Moderate to Severe | 0
  Severe to Uninfected | 0
  Severe to Mild | 0
  Severe to Moderate | 0
  Severe to Severe | 0

16. Secondary Outcome: Need for Surgery, Hospitalisation and Non-Study Antibiotic Therapy for Diabetic Foot Infection During Study (in ITT Population)
Description: Results in relation to the need for surgery, hospitalization, new and/or additional non-study antibiotic therapy for failure of initial oral therapy at End of Treatment/Early Termination.
Time Frame: End of Treatment/Early Termination Visit; 7±1, 14±1, 21±1 or 28±1 days after Baseline (Day 1)
Population: Number at the End of Treatment/Early Termination Visit, ITT population
Measure: Number; unit: participants
Arm/Group | Nemonoxacin
Number analyzed (Participants) | 32
participants
  Surgery Required for DFI During Study | 1
  Hospitalisation Required for DFI During Study | 1
  New or Additional Antibiotic Therapy Required | 3

17. Secondary Outcome: Need for Surgery, Hospitalisation and Non-Study Antibiotic Therapy for Diabetic Foot Infection During Study (in ITT Population)
Description: Results in relation to the need for surgery, hospitalization, new and/or additional non-study antibiotic therapy for failure of initial oral therapy at Test of Cure.
Time Frame: Test of Cure Visit, 12±2 days after End of Treatment Visit/Early Termination
Population: Number at Test of Cure Visit, ITT population
Measure: Number; unit: participants
Arm/Group | Nemonoxacin
Number analyzed (Participants) | 30
participants
  Surgery Required for DFI During Study | 1
  Hospitalisation Required for DFI During Study | 1
  New or Additional Antibiotic Therapy Required | 3

18. Secondary Outcome: Need for Surgery, Hospitalisation and Non-Study Antibiotic Therapy for Diabetic Foot Infection During Study (in PP Population)
Description: as for outcome 16
Time Frame: End of Treatment/Early Termination Visit; 7±1, 14±1, 21±1 or 28±1 days after Baseline (Day 1)
Measure: Number; unit: participants
Arm/Group | Nemonoxacin
Number analyzed (Participants) | 20
participants
  Surgery Required for DFI During Study | 0
  Hospitalisation Required for DFI During Study | 0
  New or Additional Antibiotic Therapy Required | 0

19. Secondary Outcome: Need for Surgery, Hospitalisation and Non-Study Antibiotic Therapy for Diabetic Foot Infection During Study (in PP Population)
Description: as for outcome 17
Time Frame: Test of Cure Visit, 12±2 days after End of Treatment Visit/Early Termination
Measure: Number; unit: participants
Arm/Group | Nemonoxacin
Number analyzed (Participants) | 20
participants
  Surgery Required for DFI During Study | 0
  Hospitalisation Required for DFI During Study | 0
  New or Additional Antibiotic Therapy Required | 1

ADVERSE EVENTS:
Time Frame: Study period (Visit 1 to Test of Cure)
Description: At each visit, the Investigator will determine whether any adverse events have occurred. The patients will be questioned in a general way and no specific symptoms will be suggested. None of the SAEs were considered related to study drug. No patient died during the study period.
Arm/Group | Nemonoxacin
Serious Adverse Events (participants affected / at risk) | 5/38
Other Adverse Events (participants affected / at risk) | 21/38
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Nemonoxacin (N=38)
GANGRENE (Infections and infestations) | 2
ABSCESS LIMB (Infections and infestations) | 1
OSTEOMYELITIS (Infections and infestations) | 1
BLOOD GLUCOSE INCREASED (Investigations) | 1
BLOOD PRESSURE INCREASED (Investigations) | 1
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Nemonoxacin (N=38)
OSTEOMYELITIS (Infections and infestations) | 3
CELLULITIS (Infections and infestations) | 2
GANGRENE (Infections and infestations) | 2
ABSCESS LIMB (Infections and infestations) | 1
INFECTION (Infections and infestations) | 1
CONSTIPATION (Gastrointestinal disorders) | 2
DIARRHOEA (Gastrointestinal disorders) | 2
VOMITING (Gastrointestinal disorders) | 1
BLOOD GLUCOSE INCREASED (Investigations) | 3
BLOOD ALBUMIN DECREASED (Investigations) | 1
BLOOD PRESSURE INCREASED (Investigations) | 1
BLOOD UREA INCREASED (Investigations) | 1
CREATININE RENAL CLEARANCE DECREASED (Investigations) | 1
ELECTROCARDIOGRAM QT PROLONGED (Investigations) | 1
PAIN IN EXTREMITY (Musculoskeletal and connective tissue disorders) | 2
MYALGIA (Musculoskeletal and connective tissue disorders) | 1
NECK PAIN (Musculoskeletal and connective tissue disorders) | 1
OSTEITIS (Musculoskeletal and connective tissue disorders) | 1
SKIN ULCER (Skin and subcutaneous tissue disorders) | 2
PRURITUS GENERALISED (Skin and subcutaneous tissue disorders) | 1
RASH PRURITIC (Skin and subcutaneous tissue disorders) | 1
SKIN FISSURES (Skin and subcutaneous tissue disorders) | 1
SWELLING FACE (Skin and subcutaneous tissue disorders) | 1
HEADACHE (Nervous system disorders) | 3
EPISTAXIS (Respiratory, thoracic and mediastinal disorders) | 1
INCREASED UPPER AIRWAY SECRETION (Respiratory, thoracic and mediastinal disorders) | 1
THROAT TIGHTNESS (Respiratory, thoracic and mediastinal disorders) | 1
DIABETIC RETINOPATHY (Eye disorders) | 1
EYE PAIN (Eye disorders) | 1
HYPERGLYCAEMIA (Metabolism and nutrition disorders) | 1
HYPOGLYCAEMIA (Metabolism and nutrition disorders) | 1
ANAEMIA (Blood and lymphatic system disorders) | 1
FOOT FRACTURE (Injury, poisoning and procedural complications) | 1
PERSONALITY CHANGE (Psychiatric disorders) | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
PI needs to inform sponsor and asks for permission before he/she discusses or publishes trial results after the trial is completed.